CLINICAL TRIAL: NCT06652698
Title: Early Supplementation for Cow's Milk Allergy Prevention in Breastfed Infants in Poland (ESCAPE-PL): a Protocol for Randomised Controlled Trial
Brief Title: Early Supplementation for Cow's Milk Allergy Prevention
Acronym: ESCAPE-PL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ABM30
Record Dates: First submitted 2024-07-23; First posted 2024-10-22 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Food Allergy; Cow's Milk Allergy
MeSH Terms: conditions — Food Hypersensitivity; Milk Hypersensitivity | interventions — CMF regimen; 2-Acetylaminofluorene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CMF (Experimental)
  Interventions: Other: Cow's milk formula [CMF]
- AAF (Experimental)
  Interventions: Other: Amino-acid formula [AAF]
- DHM (Experimental)
  Interventions: Other: Donor human milk [DHM]
- DHM-P (Experimental)
  Interventions: Other: High-pressure processed "pascalized" donor human milk [DHM-P]

INTERVENTIONS:
Other: Cow's milk formula [CMF] — At least 10 ml daily of cow's milk formula (Bebiko 1 NUTRIFlor Expert®, Nutricia; formula with galactooligosaccharides and without probiotics); and if additional supplementation will be needed (i.e., insufficient, partial, or discontinuation of breastfeeding), the randomly assigned nutritional intervention until the end of 4 months of age will be provided.
  Arms: CMF
Other: Amino-acid formula [AAF] — At least 10 ml daily of amino-acid formula (Nutramigen Pureamino®, Reckitt Benckiser Group PLC); and if additional supplementation will be needed (i.e., insufficient, partial, or discontinuation of breastfeeding), the randomly assigned nutritional intervention until the end of 4 months of age will be provided.
  Arms: AAF
Other: Donor human milk [DHM] — At least 10 ml daily of donor human milk; and if additional supplementation will be needed (i.e., insufficient, partial, or discontinuation of breastfeeding), the randomly assigned nutritional intervention until the end of 4 months of age will be provided.
  Arms: DHM
Other: High-pressure processed "pascalized" donor human milk [DHM-P] — At least 10 ml daily of high-pressure processed "pascalized" donor human milk; and if additional supplementation will be needed (i.e., insufficient, partial, or discontinuation of breastfeeding), the randomly assigned nutritional intervention until the end of 4 months of age will be provided.
  Arms: DHM-P

SUMMARY:
Cow's milk allergy (CMA) is a common food allergy in infants and young children that can have a significant impact on the individual and their family due to dietary restrictions, risk of nutritional deficiencies, social limitations, and decreased quality of life. It also represents a financial burden for families and healthcare resources.

There is an ongoing debate about the significance of early exposure to cow's milk proteins within hours or days after birth and its relationship to the risk of developing CMA later in life. Current recommendations for early introduction of cow's milk proteins in infants who cannot be breastfed vary and are inconsistent due to a lack of clear evidence. This knowledge gap underscores the need for further research to provide a definitive understanding of the relationship between early exposure to cow's milk proteins and the development of CMA, which will ultimately inform evidence-based prevention strategies to improve the health and well-being of affected individuals and their families.

This trial aims to investigate whether early supplementation with various nutritional interventions (cow's milk formula [CMF], amino acids formula [AAF], donor human milk [DHM], or high-pressure processed "pascalized" donor human milk [DHM-P]) could serve as an effective strategy for the primary prevention of CMA in breastfed neonates.

This study is an open-label randomized, controlled, head-to-head trial with four parallel arms and allocation 1:1:1:1.

ELIGIBILITY:
Inclusion criteria:

1. Healthy newborns of mothers who express the intention to exclusively breastfeed for first 6 months of infant's life
2. Full-term infants (defined as gestational age of at least 37 weeks)
3. Infant birth weight at least 2500 g and ≤ 4500 g
4. Age at enrolment <24 h of life
5. Regardless of any atopic condition in parents
6. Written informed consent of the caregiver

Exclusion criteria:

1. Infants of parents who intend to partially or fully formula feed
2. Serious congenital anomalies or any other medical condition that would preclude the consumption of any of the study formulas, or interfere with nutrition or growth
3. Contradictions to exclusive breastfeeding
4. Multiple pregnancy

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
A cumulative incidence of cow's milk allergy confirmed by open oral food challenge | At 4-6 and 12 months of age

SECONDARY OUTCOMES:
A cumulative incidence of sensitization to cow's milk protein (cut-off levels for specific IgE level ≥0.35 allergen units [UA/mL] and ≥3 mm of wheal size in the skin prick test against cow's milk | at 6 and 12 months of age
A point prevalence of cow's milk allergy confirmed by open oral food challenge | at 4-6, and 12 months of age
An incidence of sensitization to cow's milk protein (cut-off levels for specific IgE level ≥0.35 allergen units [UA/mL] against cow's milk) | at 4-6, and 12 months of age
In a subgroup of children with confirmed cow's milk allergy, the percentage of children with tolerance acquisition to cow's milk | at 9 and/or 12 months
  Tolerance acquisition to cow's milk will be assessed by subsequent OFC with baked milk (in the form of biscuit or muffin); if baked milk is tolerated, the assessment of tolerance acquisition will be continued with the use of milk ladder.
Percentage of children who received a full 3-day nutritional supplementation (3x10 ml according to the randomization) and then were exclusively or predominantly breastfed until 4 months of age | Up to 4 month of age
A total score in the Cow's Milk-related Symptom Score (CoMiSS) | at 4-6 and 12 months of age
  The total CoMiSS score ranges from 0 to 33, a score of ≥10 indicates CMA.
Percentage of children exclusively breastfed | at 4 and 6 months of age
Percentage of children with mixed feeding | at 4 and 6 months of age
Change in Body Mass Index (BMI)-for-age z-score | at 4, 6 and 12 months of age
  weight and length will be checked each month in a telephone interview or parental report, or during follow-up visit assessed by study physician; change in mean value will be assessed between baseline and each time point
Change in length-for-age z-score | at 4, 6 and 12 months of age
  length will be checked each month in a telephone interview or parental report, or during follow-up visit assessed by study physician; change in mean value will be assessed between baseline and each time point
Adverse events related to the nutritional intervention (according to the randomization) | up to 12 months of age
  defined as any harmful events that may occur during the trial; the process of decision whether an adverse event is related to the intervention (attribution) will be made by the non-blinded principal investigator
A cumulative incidence of atopic dermatitis (defined as meeting the UK Working Party diagnostic Criteria) | at 6 and 12 months of age
A cumulative incidence of allergic rhinitis (confirmed by study physician) | at 6 and 12 months of age
A cumulative incidence of feeding difficulties who will be screened with The Montreal Children's Hospital Feeding Scale (MCH-FS scale) | at 6 and 12 months of age
  Total score range from 14 to 98, score of 46 or higher indicates feeding difficulties.
Human milk energy value (kcal/100 mL) | at 4-14 days postpartum and 6 months of age
Total and true protein concentrations in human milk samples (g/100 mL) | at 4-14 days postpartum and 6 months of age
Fat concentration in human milk samples (g/100 mL) | at 4-14 days postpartum and 6 months of age
Lactose concentration in human milk samples (g/100 mL) | at 4-14 days postpartum and 6 months of age
Dry mass content g/100 mL | at 4-14 days postpartum and 6 months of age
IgA-anty CMA concentration in human milk samples (pg/mL) | at 4-14 days postpartum
IL-1B, IL-6, IL-10, and TGF-beta concentrations in human milk samples (pg/mL) | at 4-14 days postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Horvath, Assoc Prof, MD, Study Chair — Medical University of Warsaw; Aleksandra Wesołowska, Assoc Prof, Principal Investigator — Medical University of Warsaw; Hanna Szajewska, Prof, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The anonymized datasets used and/or generated during this study will be made available from a corresponding author on reasonable request, after the publication of results, no later than 3 years from the completion of data analysis.
Supporting Information: CSR
Time Frame: After the publication of results, no later than 3 years from the completion of data analysis.
Access Criteria: The anonymized datasets used and/or gener.ated during this study will be made available from a corresponding author on reasonable request

REFERENCES:
- [Derived] Horvath A, Wesolowska A, Strozyk A, Bzikowska-Jura A, Ambrozej D, Dumycz K, Feleszko W, Szajewska H. Early supplementation for cow's milk allergy prevention in breastfed infants in Poland (ESCAPE-PL): a protocol for randomised controlled trial. BMJ Open. 2025 Aug 5;15(8):e096217. doi: 10.1136/bmjopen-2024-096217. PMID 40764079